CLINICAL TRIAL: NCT03694899
Title: The Excess Opioid Disposal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., Chief, Section of General Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D19001
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one (Experimental): acetaminophen 650 mg three times/day ibuprofen 600 mg three times/day opioid dose based on use in hospital day prior to discharge
  Interventions: Behavioral: phone contact

INTERVENTIONS:
Behavioral: phone contact — patients will be called prior to their outpatient appointment

SUMMARY:
This study is designed to test the hypothesis that providing information to patients about excess opioid disposal, calling patients prior to their outpatient post-operative surgical appointment and providing a convenient drop box for opioid disposal will increase rates of FDA compliant disposal.

DETAILED DESCRIPTION:
It is hypothesized that:

1. By providing pre-operative patient education, a drop-box in a convenient location (the hospital pharmacy near the surgical outpatient clinic) and a reminder phone call prior to the post-operative clinic appointment, an increase in FDA-compliant unused opioid disposal rates to at least 40% will be seen.
2. The investigator's guideline for opioid prescribing after operations that require an inpatient admission which the investigator established for general surgical procedures will satisfy the opioid requirements of at least 85% of patients undergoing a variety of operations from differing specialties.
3. The utilization of guideline opioid prescribing and FDA-compliant unused opioid disposal will decrease the percentage of patients who are taking opioids at 6 months and 1 year after their surgery to less than 1%.

The primary objective is to determine the effect of pre-operative patient education, a drop-box in the hospital pharmacy and a reminder phone call on the proportion of patients who dispose of unused opioids using a FDA-compliant method.

Secondary objectives include:

1. Determine in a prospective study whether our guideline for opioid prescribing after surgery which requires inpatient admission fulfills the opioid requirements of at least 85% of patients undergoing a variety of operations.
2. Determining the effect of guideline opioid prescribing and FDA-compliant unused opioid disposal on the proportion of patients who are on opioids 6 months and 1 year after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having surgery with expected duration of admission of 2 days or more

Exclusion Criteria:

* Allergies to opioids
* Allergy or contra-indication to short term acetaminophen or ibuprofen
* Chronic opioid use
* History of opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
opioid disposal rate | 1 year
  % of patients that dispose of excess opioids in an FDA compliant manner

SECONDARY OUTCOMES:
Does guideline predict opioid needs | 6 months
  1.Determine in a prospective study whether our guideline for opioid prescribing after surgery which requires inpatient admission fulfills the opioid requirements of at least 85% of patients undergoing a variety of operations.
effect on long term opioid usage | 1 year
  Determining the effect of guideline opioid prescribing and FDA-compliant unused opioid disposal on the proportion of patients who are on opioids 6 months and 1 year after their surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porter ED, Bessen SY, Molloy IB, Kelly JL, Ramkumar N, Phillips JD, Loehrer AP, Wilson MZ, Hasson RM, Ivatury SJ, Henkin JR, Barth RJ Jr. Guidelines for Patient-CenteredOpioid Prescribing and Optimal FDA-Compliant Disposal of Excess Pills after Inpatient Operation: Prospective Clinical Trial. J Am Coll Surg. 2021 Jun;232(6):823-835.e2. doi: 10.1016/j.jamcollsurg.2020.12.057. Epub 2021 Feb 25. PMID 33640521